CLINICAL TRIAL: NCT03414775
Title: Influences of High-fiber, Organic Whole-food Formula on the Gut Microbiome in Critically Ill Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Rajesh Aneja, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY19080289
Record Dates: First submitted 2018-01-22; First posted 2018-01-30 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Critical Illness; Dysbiosis; Pediatric ALL
Keywords: microbiome; gastrointestinal microbiome; pediatrics; critical illness
MeSH Terms: conditions — Critical Illness; Dysbiosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Critically-ill children who are medically stable and ready for enteral tube feeds will be randomized to receive either Pediasure or Nourish. Nutritional needs will be calculated per previously established standards at our institution and performed in conjunction with trained dieticians and nutritionists.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pediasure (Active Comparator): Patients assigned to this arm will receive Pediasure
  Interventions: Other: Pediasure
- Nourish (Active Comparator): Patients assigned to this arm will receive Nourish
  Interventions: Other: Nourish

INTERVENTIONS:
Other: Nourish — The effects of Nourish on the gastrointestinal microbiome will be compared to the the effects of Pediasure on the gastrointestinal microbiome
  Arms: Nourish
Other: Pediasure — The effects of Nourish on the gastrointestinal microbiome will be compared to the the effects of Pediasure on the gastrointestinal microbiome
  Arms: Pediasure

SUMMARY:
This study evaluates the effects of either Pediasure or Nourish formulas on the gastrointestinal microbiome in critically-ill children. Patients will be randomized to received either Pediasure or Nourish.

DETAILED DESCRIPTION:
The gastrointestinal microbiome has been shown to be altered in critically-ill children such that there is a larger shift toward pathogenic bacteria. Previous studies have shown that probiotics, fecal transplants, antibiotic decontamination, and dietary interventions can shift the gastrointestinal microbiome toward a metabolically favorable microbiome profile and be associated with improvements in disease burden.

This study will randomize critically-ill children who are stable enough for enteral tube feedings to receive either Pediasure or Nourish. Pediasure is a commercially-made formula that is used commonly in pediatric patients. Nourish is an organic, whole-food formula with a high fiber content. High-fiber diets have been correlated with metabolically favorable microbiome profiles. This study will look at the microbiome before and after initiation of enteral tube feedings to determine if either formula is associated with a shift in the microbiome toward a favorable profile.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the pediatric intensive care unit
* Age 1-17 years old
* Previously placed enteric tube designed for enteric feeding

Exclusion Criteria:

* Vasoactive medication use
* History of allergies or intolerances to either Pediasure or Nourish
* Whey allergy or intolerance
* Gluten sensitivity or intolerance
* Medical condition that necessitate the use of specific formulas and/or nutritional needs (e.g. epilepsy requiring ketogenic diet, genetic metabolic dysfunction with specific formula requirements)

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Changes to the gastrointestinal microbiome | Prior to initiation of enteral tube feeds then on day 1, day 5-7, and day 14 of feedings
  Fecal samples will be collected for bacterial 16s rRNA gene sequencing and analysis
Changes to the gastrointestinal microbiome | Prior to initiation of enteral tube feeds then on day 1, day 5-7, and day 14 of feedings
  Salivary samples will be collected for bacterial 16s rRNA gene sequencing and analysis

SECONDARY OUTCOMES:
Concentration of short-chain fatty acids | Prior to initiation of enteral tube feeds then on day 1, day 5-7, and day 14 of feedings
  Fecal samples will be analyzed by gas chromatography

CONTACTS AND LOCATIONS:
Overall Officials: Raj Aneja, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No